CLINICAL TRIAL: NCT07108413
Title: Study Protocol to Investigate the Effect of a Novel Aerobic Exercise Intervention With Integrated Cognitive Training, Active4Brain, on Cognition, Neurophysiology, and Neuroprotective Markers in Older Adults
Brief Title: Study of the Cognitive and Neurophysiological Effects of the Activ4Brain Program for Older Adults
Acronym: Activ4Brain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Maria Ribeiro, Principal Investigator, University of Coimbra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Activ4Brain
Record Dates: First submitted 2025-07-07; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Older People
Keywords: Aerobic exercise; Cognitive training; Age-related cognitive decline; Electroencephalography (EEG); Immune function biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Activ4Brain Group (Experimental): Participants in this group perform the Activ4Brain program during 3 months
  Interventions: Behavioral: Activ4Brain Program
- Aerobic exercise group (Active Comparator): Participants in this group perform an Aerobic Exercise program during 3 months
  Interventions: Behavioral: Aerobic Exercise Program
- Control group (No Intervention): Participants in this group receive no intervention during the study and are instructed to carry on their daily routines.

INTERVENTIONS:
Behavioral: Activ4Brain Program — The Activ4Brain Program consists of 24 sessions, twice a week for 3 months. Participants engage in 50 min exercise sessions of moderate intensity (60-80% of maximal heart rate) including 5 min warm-up, 40 min aerobic exercises, and 5 min cool-down. The warm-up period includes similar body movements as the main part of the exercise and dynamic stretching while the cool down period consists of static stretching. The main part of the exercise session is divided in four blocks. Each block consists of 5 min aerobic exercises and 5 min of cognitive training. Participants are instructed to keep moving, marching in place, while performing the cognitive training tasks to maintain the increased heart rate. Each group class is composed of four participants with as must as possible a narrow age range given the participants' schedule convenience.
  Arms: Activ4Brain Group
Behavioral: Aerobic Exercise Program — The Aerobic Exercise Program consists of 24 sessions, twice a week for 3 months. Participants engage in 50 min exercise sessions of moderate intensity (60-80% of maximal heart rate) including 5 min warm-up, 40 min aerobic exercises, and 5 min cool-down. The warm-up period includes similar body movements as the main part of the exercise and dynamic stretching while the cool down period consists of static stretching. The main part of the exercise session consists of a sequence of four different 5 min blocks of aerobic exercise repeated twice. Each block consists of a combination of three different rhythmic movements. Each group class is composed of four participants.
  Arms: Aerobic exercise group

SUMMARY:
This study aims to examine the cognitive, neuronal, and physical effects of the Activ4Brain program in older men and women between 55 and 75 years of age. The program Activ4Brain consists of 24 sessions of aerobic exercise classes (twice a week over 3 months) that include computerized games designed to train cognition. Participants are tested before and after the 3-months intervention. Researchers will study changes in cognitive function, brain and body physiological activity, and inflammation and neuroprotective markers in 3 groups of participants: the Activ4Brain group that engages in the Activ4Brain program, an active control group that engages in aerobic exercise classes and a passive control group that does not engage in any intervention.

This study aims to answer the following questions.

* Does the program Activ4Brain improve cognition in cognitively healthy older adults?
* Does the program Activ4Brain change brain function and body physiology in cognitively healthy older adults?

DETAILED DESCRIPTION:
Cognitive training and physical exercise hold the potential to be successful non-pharmacological treatments for age-related cognitive decline and dementia. However, existing interventions show little to no benefit for preventing or delaying cognitive decline, highlighting the need to develop alternative tools. With this in mind, the Activ4Brain program was designed as a non-pharmacological strategy to reduce the impact of age-related cognitive decline. The Activ4Brain program consists of group aerobic exercise classes where computerized games targeting different cognitive domains are applied during the session to potentiate the effect of physical exercise on cognition. This study investigates the impact of this novel program on cognitive and brain function.

The primary objective of this study is:

• Evaluation of the efficacy of the Activ4Brain program in improving cognition in older people

Secondary objectives are:

* Evaluation of the impact of the Activ4Brain program on brain and autonomic function and physical health markers
* Evaluation of participants' adherence and retention through attendance rates across all intervention sessions and participation trends over time
* Evaluation of the feasibility of the Activ4Brain program including its acceptability, accessibility, and usability.

ELIGIBILITY:
Inclusion Criteria:

• Men and women between 55 and 75 years of age

Exclusion Criteria:

* Presence of contraindications for physical exercise screened with the Physical Activity Readiness Questionnaire (PAR-Q)
* Presence of objective cognitive impairment screened with the Addenbroke's Cognitive Examination - Revised, which also incorporates the Mini Mental State Examination, providing a double score
* Presence of high fall risk screened with the Timed Up and Go test (TUG)
* Presence of severe neurological or psychiatric conditions

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Executive Function - Multitasking test from the CANTAB Research Connect | From one month before the 3-months intervention up to one month after the end of the intervention.
  Executive function will be assessed with the Multitasking test from the CANTAB Research Connect (Cambridge Cognition Ltd) - 3-months score change in MTT Multitasking cost (median). The score is calculated by subtracting the median latency of response during single task block(s) from the median latency of response during multitasking block(s). A positive score indicates that the subject responds more slowly during multitasking blocks and indicates a higher cost of managing multiple sources of information. Lower values are associated with better executive function.
Change from Baseline in Working Memory - Spatial Working Memory (SWM) test from the CANTAB Research Connect | From one month before the 3-months intervention up to one month after the end of the intervention.
  Working memory will be assessed with the Spatial Working Memory (SWM) test from the CANTAB Research Connect (Cambridge Cognition Ltd)- 3-months score change in SWM Between Errors: the number of times the subject incorrectly revisits a box in which a token has previously been found. Lower values are associated with better working memory abilities.
Change from Baseline in Episodic Memory - Auditory Verbal Learning Test | From one month before the 3-months intervention up to one month after the end of the intervention.
  Auditory Verbal Learning Test (AVLT) - 3-months score change in Total Learning: the sum of words remembered across Trial 1 through Trial 5. Higher values represent better memory abilities.
Change from Baseline in Sustained Attention - Rapid Visual Information Processing test from the CANTAB Research Connect | From one month before the 3-months intervention up to one month after the end of the intervention.
  Sustained attention will be assessed with the Rapid Visual Information Processing test from the CANTAB Research Connect (Cambridge Cognition Ltd) - 3-months score changes in RVPA (subject's sensitivity to the target sequence). Higher values represent better sustained attention scores.
Change from Baseline in Processing Speed - Rapid Visual Information Processing test from the CANTAB Research Connect | From one month before the 3-months intervention up to one month after the end of the intervention.
  Processing speed will be assessed with the Rapid Visual Information Processing test from the CANTAB Research Connect (Cambridge Cognition Ltd) - 3-months score change in RVP Median Response Latency (median response latency on correct trials). Lower values represent faster processing speed.
Change from Baseline in Processing Speed - Multitasking test from the CANTAB Research Connect | From one month before the 3-months intervention up to one month after the end of the intervention.
  Processing speed will be assessed with the Multitasking test from the CANTAB Research Connect (Cambridge Cognition Ltd) - 3-months score change in MTT Incongruency cost (difference between the median response latency on the congruent versus incongruent trials). A lower incongruency cost indicates that the subject processes conflicting information faster.

SECONDARY OUTCOMES:
1. Change from Baseline in the Amplitude of Event-Related Potentials Evoked during a Reinforcement Learning Task | From one month before the 3-months intervention up to one month after the end of the intervention.
  Change in event-related potentials evoked during a reinforcement learning task are assessed using amplitude (microV) measures of event-related potentials recorded using a 64-channel Neuroscan system (Compumedics EUROPE GmbH) with scalp electrodes placed according to the International 10-20 electrode system (500 Hz sampling rate).
Change from Baseline in Amplitude of Pupil Responses during a Reinforcement Learning Task. | From one month before the 3-months intervention up to one month after the end of the intervention.
  Amplitude of task-related pupil responses during cognitive task performance are assessed using pupil size data obtained with an eye tracking system recorded during a reinforcement learning task. Amplitude of pupil responses are measured in normalized units as percentage of the mean pupil size for each participant.
Change from Baseline in the Amplitude of Task-Related Heart Rate Responses Evoked during a Reinforcement Learning Task. | From one month before the 3-months intervention up to one month after the end of the intervention.
  Task-related heart rate responses that occur during a reinforcement learning task are calculated from the electrocardiogram recorded with bipolar electrodes attached to the participants' chest. Task-related heart rate responses are measured as changes in cardiac interbeat-interval associated with task events.
Change from Baseline in Heart Rate Variability during Rest - time domain measures | From one month before the 3-months intervention up to one month after the end of the intervention.
  3-month change in Mean RR (ms), SDNN (ms), RMSSD (ms).
Change from Baseline in Heart Rate Variability during Rest - frequency domain measures | From one month before the 3-months intervention up to one month after the end of the intervention.
  3-month change in VLF (ms^2), LF (ms^2), and HF (ms^2).
Change from Baseline in the Concentration of Blood Plasma Levels of Inflammatory Biomarkers | From one month before the 3-months intervention up to one month after the end of the intervention.
  Changes in concentration of inflammatory blood biomarkers are assessed in blood samples collected from venous blood (15 ml) in a fasting state, in the morning. Plasma samples will be quantified by ELISA for Interleukin (IL)-6 (pg/ml), IL-1β (pg/ml), Tumor Necrosis Factor (TNF)-α (pg/ml), Interferon(IFN) -γ (pg/ml), IL-17, (pg/ml).
Change from Baseline in the Concentration of Blood Plasma Levels of Anti-Inflammatory Biomarkers | From one month before the 3-months intervention up to one month after the end of the intervention.
  Changes in concentration of anti-inflammatory biomarkers are assessed in blood samples collected from venous blood (15 ml) in fasting state, in the morning. Plasma samples will be quantified by ELISA (Thermofisher, UK) for IL-1Ra (pg/ml), IL-10 (pg/ml).
Change from Baseline in the Concentration of Vascular Endothelial Growth Factor-D (VEGF-D) Blood Serum Levels | From one month before the 3-months intervention up to one month after the end of the intervention.
  Changes in concentration of Vascular Endothelial Growth Factor-D (VEGF-D) are assessed in blood samples collected from venous blood (15 ml) in fasting state, in the morning. Serum samples will be quantified by ELISA for VEGF-D (pg/ml).
Change from Baseline in the Concentration of Insulin-Like Growth Factor 1 (IGF-1) Blood Serum Levels | From one month before the 3-months intervention up to one month after the end of the intervention.
  Changes in concentration of Insulin-Like Growth Factor 1 (IGF-1) are assessed in blood samples collected from venous blood (15 ml) in fasting state, in the morning. Serum samples will be quantified by ELISA for IGF-1 (ng/ml).
Change from Baseline in the Concentration of Neurotrophic Factors Blood Serum Levels | From one month before the 3-months intervention up to one month after the end of the intervention.
  Changes in concentration of Neurotrophic Factors are assessed in blood samples collected from venous blood (15 ml) in fasting state, in the morning. Serum samples will be quantified by ELISA for Brain-Derived Neurotrophic Factor (BDNF)(ng/ml) and Glial cell line-Derived Neurotrophic Factor (GDNF)(ng/ml).
Change from Baseline in the Concentration of Irisin Blood Serum Levels | From one month before the 3-months intervention up to one month after the end of the intervention.
  Changes in concentration of Irisin (pg/ml) are assessed in blood samples collected from venous blood (15 ml) in fasting state, in the morning. Serum samples will be quantified by ELISA.
Feasibility Outcomes: Adherence to the Intervention Protocols | One month after the intervention
  Adherence to the intervention protocols is assessed by evaluating the attendance rates (percentage of intervention sessions that were attended per participant).
Feasibility Outcomes: Retention | One month after the intervention
  Retention is quantified at the end of the study from dropout data: percentage of participants that terminated the intervention and completed the follow-up testing procedures in each group.
Feasibility Outcomes: Average Group Scores in Acceptability Scale | From the end of the intervention up to one month after the intervention.
  Program acceptability measured with custom made acceptability scale applied to the Activ4Brain and Aerobic Exercise groups. The scale is composed of 4 items and the responses are recorded on a scale ranging from 1 to 5 where larger values are associated with higher acceptability. The acceptability score is calculated as the average score of the 4 items.
Feasibility Outcomes: Average Group Scores in the System Usability Scale (SUS) | From the end of the intervention up to one month after the intervention.
  Usability of the Activ4Brain cognitive training system measured with the System Usability Scale (SUS) applied to the Activ4Brain group. SUS is composed of 10 items, each measured on a scale from 1 to 5, and yields a single number representing a composite measure of the overall usability of the system being studied. Each item's score contribution ranges from 0 to 4. For items 1, 3, 5, 7, and 9 the score contribution is the scale position minus 1. For items 2, 4, 6, 8 and 10, the contribution is 5 minus the scale position. The sum of the scores is then multiplied by 2.5 to obtain the overall value of System Usability. SUS scores have a range of 0 to 100.

OTHER OUTCOMES:
Change from Baseline in Peak Oxygen Consumption (VO2) | From one month before the 3-months intervention up to one month after the end of the intervention.
  Peak oxygen uptake capacity (VO2 peak) measured in mL/min/Kg, with a submaximal incremental cycle ergometry test (Lode- Excalibur, Netherlands), before and after the intervention. Following a warm-up period, participants started the testing phase with an initial load of 50 watts for women and 75 watts for men33. The load is increased by 25 watts at every three-minute intervals. The test continues at 60-70 rpm and is completed once participants achieve 85% of their predicted maximal heart rate, as determined by the Tanaka Formula.
Change from Baseline in Body Composition | From one month before the 3-months intervention up to one month after the end of the intervention.
  Changes in body composition is measured for total body mass (kg), fat mass (kg), fat free mass (kg) by bioimpedance.
Change from Baseline in Body Mass Index (BMI) | From one month before the 3-months intervention up to one month after the end of the intervention.
  3-months change in body mass index: weight and height will be combined to calculate BMI in kg/m^2).
Change from Baseline in Phase Angle | From one month before the 3-months intervention up to one month after the end of the intervention.
  3-months change in Phase Angle (°) calculated automatically by the Inbody 770 device (Biospace) with following formula (°) = (reactance/resistance) × (180/π).

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Ribeiro, PhD, Principal Investigator — CIBIT-ICNAS, University of Coimbra, Portugal
Locations (1):
- University of Coimbra, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: social media page of the Activ4Brain program — https://www.facebook.com/profile.php?id=61569014774373